CLINICAL TRIAL: NCT01680757
Title: Multicenter Registry of Permanent Ligation Approximation Closure Exclusion of the Left Atrial Appendage in Patients With Atrial Fibrillation III (PLACE III)
Brief Title: Study of Left Atrial Appendage Closure in Patients With Atrial Fibrillation - III
Acronym: PLACE III
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: This study has been withdrawn prior to enrollment
Sponsor: University of California, San Francisco (Other)
Collaborators: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: RS-001 PLACE III
Record Dates: First submitted 2012-08-28; First posted 2012-09-07 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Atrial Fibrillation
Keywords: Left Atrial Appendage; LARIAT; atrial fibrillation; contraindication to oral anticoagulation therapy
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LAA exclusion with LARIAT & Accessories (Experimental): Permanent exclusion of the LAA using the LARIAT Suture Delivery Device and Accessories
  Interventions: Device: LARIAT Suture Delivery Device and Accessories

INTERVENTIONS:
Device: LARIAT Suture Delivery Device and Accessories
  Other Names: LARIATTM Suture Delivery Device; ENDOCATH Occlusion Balloon; SOFTIPTM Guide Cannula; FINDRWIRZ Guide Wire System; SURECUT Suture Cutter; TENSURE Suture Puller

SUMMARY:
This study is a prospective, multicenter, non-randomized trial of a stand-alone procedure for left atrial appendage exclusion in patients with atrial fibrillation at risk for embolic events who are contraindicated for or intolerant of oral anticoagulation therapy. This study will enroll 100 participant, who will receive the LAA ligation study treatment. The objective of this registry is to assess the effectiveness of permanent exclusion of the LAA using the LARIAT Suture Delivery Device and Accessories in patients unable to be treated with standard anticoagulation therapy. The results of the study will be used to assess outcomes within the first year, post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 21 years
2. Diagnosed non-valvular atrial fibrillation
3. Current CHADS2 score > 2
4. Currently contraindicated to or intolerant of standard anticoagulation therapy (i.e., warfarin, dabigatran, apixaban, and rivaroxaban) due to at least one of the following: history of bleeding or high risk of bleeding; labile INR level (While on anticoagulation therapy, participant had INR results "out of therapeutic range" > 40% of the time, over a minimum period of 2 months.); non-compliant, unwilling to take, or anticoagulant failure (e.g., TIA or stroke while on anticoagulant therapy).
5. Life expectancy of at least 1 year
6. Willing and able to return and comply with scheduled follow up visits
7. Willing and able to provide written informed consent

Exclusion Criteria:

1. Prior cardiac surgery involving opening of pericardium (e.g., CABG, heart transplantation, valve surgery)
2. Prosthetic heart valve or ring in any position
3. Current NYHA Class IV heart failure symptoms
4. Current right heart failure
5. Myocardial infarction within last 3 months
6. Unstable angina within last 3 months
7. Current cardiogenic shock or hemodynamic instability
8. Current symptomatic carotid disease
9. Need for an intra-aortic balloon pump or intravenous inotropes
10. Embolic stroke within the last 30 days
11. Transient ischemic attack (TIA) within the last 30 days
12. Current diagnosis of active systemic infection
13. eGFR < 60 mL/min/1.73m2 within last 3 months
14. Current renal failure requiring dialysis
15. ALT or AST level > 3 times upper level of normal, indicating hepatic failure. (NOTE: normal range provided by local laboratory performing the measurement), based on most recent pre-procedure assessment (within 30 days of study treatment)
16. Current clinical evidence of cirrhosis
17. Any history of thoracic radiation
18. Current use of long term treatment with steroids, not including intermittent use of inhaled steroids for respiratory diseases
19. Diagnosed autoimmune disease known to be associated with pericarditis (i.e., specific connective tissue disorders)
20. Any history of pericarditis
21. Pectus excavatum (clinically defined by treating physician)
22. Severe scoliosis
23. Thrombocytopenia (platelet count < 100 x 109/L) based on most recent pre-procedure assessment (within 30 days of study treatment)
24. Anemia with hemoglobin concentration of < 10 g/dL based on most recent pre-procedure assessment (within 30 days of study treatment)
25. Pregnancy or desire to get pregnant within next 12 months.
26. Current enrollment in an investigation or study of a cardiovascular device or investigational drug that would interfere with this registry
27. Mental impairment or other conditions, which may not allow patient to understand the nature, significance and scope of the study
28. Any other criteria, which would make the patient unsuitable to participate in this study as determined by clinical site Principal Investigator (e.g., an uncontrolled drug and/or alcohol addiction)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Rate of complete exclusion | During 1 year follow-up.
  To assess the rate of complete exclusion of the left atrial appendage (defined as < 1 mm of communication between left appendage and atrium) measured by color duplex transesophageal echocardiography TEE).

OTHER OUTCOMES:
Rate of procedural success | Baseline
  Exploratory objectives include assessment of the rate of procedural success (defined as completion of the procedure as intended at baseline, as assessed by the clinical site Principal Investigator)
Rate of complications | During 1 year follow-up
  Exploratory objectives include assessment of the rate of complications related to the use of the LARIAT and accessories

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Marcus, MD, Principal Investigator — University of California, San Francisco
Locations (12):
- United States (10):
  - Banner Good Samaritan, Phoenix, Arizona
  - Scripps Green Hospital and Clinic, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Baptist Hospital of Miami, Miami, Florida
  - University of Kansas Hospital and Medical Center, Kansas City, Kansas
  - Columbia University Medical Center, New York, New York
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Texas Heart Institute, Houston, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - Swedish Medical Center, Seattle, Washington
- Cardiovascular Center Frankfurt, Frankfurt, Germany
- John Paul II Hospital, Krakow, Poland